CLINICAL TRIAL: NCT06604338
Title: Evaluation of Predisposing Factors for Idiopathic Recurrent Pregnancy Losses: a Study Using a Genomic and Microbiota Approach
Brief Title: Genomics and Microbiome Investigation in Cases of Recurrent Pregnancy Losses
Status: Recruiting | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20210575; 5364132100005327 (Other: Plataforma Brasil)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Pregnancy Loss(RPL)
Keywords: Miscarriage; Recurrent miscarriage; Abortion; Recurrent abortion; Genetic susceptibility; Microbiome
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Habitual; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood and cervical samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RPL group: The RPL group will include women with a history of at least two spontaneous pregnancy losses, regardless of whether they have living children, and whose etiology for the pregnancy losses was not determined by the care team's protocols.
  Interventions: Diagnostic Test: Exome test; Diagnostic Test: Microbiota analysis
- Control group: Women with at least two full-term pregnancies and no history of difficulty getting pregnant, pregnancy loss or other infertility factors will be enrolled in the control group.
  Interventions: Diagnostic Test: Microbiota analysis

INTERVENTIONS:
Diagnostic Test: Exome test — An exome will be performed on the participants of RPL group.
  Groups: RPL group
Diagnostic Test: Microbiota analysis — A cervical microbiota analysis will be performed in the RPL and control groups.

SUMMARY:
Recurrent pregnancy losses (RPL) are characterized by the occurrence of more than one spontaneous pregnancy loss. It is caused by different known factors, but about half of the cases remain without an explanation. Efforts are being done in the scientific community to solve this cases. In this study, the investigators aim to investigate genetic factors that might predispose to RPL, as well as the influence of the uterine microbiota (microorganisms that normally live in the uterus of women).

DETAILED DESCRIPTION:
Recurrent pregnancy losses (RPL) are adverse reproductive outcomes characterized by the occurrence of more than one spontaneous pregnancy loss. It is estimated that RPL occurs in 1 to 5% of couples in reproductive period and is caused by different known factors. Despite this, around half of the cases remain without a defined etiology. In this context, efforts are being done in the scientific community to elucidate idiopathic cases. Among them, robust genomic investigations, such as exome sequencing, stand out for maximizing the chances of identifying causative gene variants rather than a gene-specific approach. Another front of study to understand the factors that modulate complex etiology conditions such RPL is the characterization of the microbiota of different anatomical sites. Each human anatomical site presents a distinct microbiota selected through a long co-evolutionary process and its individual and pathological variability can lead to functional repercussions. Therefore, the aim of this study is to investigate factors predisposing to recurrent pregnancy loss through a genomic evaluation and characterization of the uterine microbiota of patients affected by RPL. To achieve this, two approaches will be conducted: a genomic approach, where the exome of women with RPL will be analyzed and compared with population genomic databases; and a etagenomic approach, where the characterization of the uterine microbiota of women with RPL will be performed and compared with that of fertile women. Using the data produced in this study, the investigators hope to be able to understand more broadly how the genome influences the predisposition to RPL and how changes in certain marker genes can lead to an increased risk for the occurrence of this reproductive condition. Furthermore, based on analyzes of the uterine microbiota, the investigators hope to be able to understand how the variability of microorganisms present in this organ acts during pregnancy, especially in cases of RPL. The results of the investigations proposed in this project will help to understand the predisposing factors to RPL and may lead to the development of new investigative approaches, such as the design of genetic panels and analyzes of the uterine microbiota, which may have an impact on the clinical management of the condition in the future.

ELIGIBILITY:
Inclusion Criteria:

* RPL group: history of at least two spontaneous pregnancy losses, regardless of whether they have living children, and whose etiology for the pregnancy losses was not determined by the care team's protocols;
* Control group: at least two full-term pregnancies and no history of difficulty getting pregnant, pregnancy loss or other infertility factors.

Exclusion Criteria:

* RPL group: less than two spontaneous pregnancy losses and those with a known cause for repeated pregnancy losses;
* Control group: N/A

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who seek the Gynecology and Obstetrics Service of the Hospital de Clínicas de Porto Alegre (HCPA) for care and investigation of causes of infertility or for exams not related to this condition will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome | At the time of enrollment
  The participants microbiome will be evaluated aiming to compare the species profile between cases and controls. The bacteria present in the microbiome will be described at the genus and species level.
Exome | At the time of enrollment
  The participants exomes will be evaluated to look for variants in specific genes, aiming to identify rare variants that will be compared with frequencies from population genomic databases. The impact of the identified variants on proteins will be assessed through in silico functional predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Rosa Fraga, PhD, Professor, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided